CLINICAL TRIAL: NCT00022256
Title: An Open-Label Phase II Trial to Evaluate the Safety and Pharmacokinetics of Motexafin Gadolinium and Cranial Irradiation in the Treatment of Newly Diagnosed Glioblastoma Multiforme
Brief Title: Motexafin Gadolinium Plus Radiation Therapy to the Brain in Treating Patients With Newly Diagnosed Glioblastoma Multiforme
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: MSKCC-01051; CDR0000068799 (Registry Identifier: PDQ (Physician Data Query)); PCI-PCYC-0206; NCI-G01-1999
Record Dates: First submitted 2001-08-10; First posted 2004-04-05 (Estimated); Last update posted 2013-06-18 (Estimated); Status verified 2013-06

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult glioblastoma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Gliosarcoma | interventions — motexafin gadolinium; Radiotherapy

INTERVENTIONS:
Drug: motexafin gadolinium
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Drugs such as motexafin gadolinium may make tumor cells more sensitive to radiation therapy.

PURPOSE: Phase II trial to study the effectiveness of motexafin gadolinium plus radiation therapy to the brain in treating patients who have newly diagnosed glioblastoma multiforme.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the safety of motexafin gadolinium and cranial irradiation, in terms of dose-limiting toxicity and clinically significant adverse events, in patients with newly diagnosed glioblastoma multiforme. II. Evaluate the pharmacokinetics of this regimen in these patients. III. Determine the survival of patients treated with this regimen. IV. Assess the activities of daily living and neurological status of patients treated with this regimen.

OUTLINE: This is a multicenter study. Patients receive motexafin gadolinium IV over 30 minutes on days 1-5 of weeks 1 and 2, and on days 1, 3, and 5 of weeks 3-6. Patients undergo cranial irradiation on days 1-5 of weeks 1-6. Treatment continues in the absence of disease progression or unacceptable toxicity. Patients undergo a neurological examination and an activities of daily living questionnaire at baseline, week 10, and during follow-up visits. Patients are followed at weeks 10 and 16 and then every 2 months thereafter.

PROJECTED ACCRUAL: A total of 20 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed glioblastoma multiforme (GBM) Grade IV astrocytoma Located supratentorially At least 2 weeks and no more than 4 weeks since prior surgery for GBM No recurrent disease

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 70-100% Life expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 50,000/mm3 Hepatic: Bilirubin no greater than 3.0 mg/dL AST and ALT no greater than 2 times upper limit of normal (ULN) Alkaline phosphatase no greater than 2 times ULN Renal: Creatinine no greater than 2.0 mg/dL Other: HIV negative No history of porphyria No glucose-6-phosphate dehydrogenase deficiency No other malignancy within the past 5 years except carcinoma in situ of the cervix or nonmelanoma skin cancer Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior antineoplastic agent for GBM No concurrent chemotherapy during and for 2 weeks after study No other concurrent antineoplastic investigational agent Endocrine therapy: Prior and concurrent corticosteroids allowed Radiotherapy: No prior radiotherapy to the brain Surgery: See Disease Characteristics Other: Concurrent anticonvulsants allowed Other concurrent cancer therapy allowed if medically necessary

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-04; Primary Completion 2003-04 (Actual); Study Completion 2003-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Josh Yamada, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States